CLINICAL TRIAL: NCT05469256
Title: Group B Streptococcus Colonization in Mother-newborn Dyads and Association With Serotype-specific Capsular Antibodies in Karachi, Pakistan.
Acronym: GBS
Status: Completed | Type: Observational
Sponsor: Aga Khan University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Emory University (Other)
Responsible Party: Principal Investigator, Dr Fyezah Jehan, Assistant Professor, Aga Khan University
Other Study IDs: 302-667
Record Dates: First submitted 2022-07-19; First posted 2022-07-21 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Group B Streptococcus (GBS) Colonization
MeSH Terms: conditions — Guillain-Barre Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Group B Streptococcus (GBS) of which there are 10 serotypes of varying invasive potential is a major cause of invasive bacterial disease in neonates and young infants. Approximately two-thirds of invasive GBS disease occurs during the first three days of life of which 75%-90% occur within 24 hours of birth in the absence of clinical interventions such as intrapartum antibiotic prophylaxis (IAP). Invasive GBS disease during the first week (Early onset disease, EOD) of life results from vertical acquisition of GBS in utero by the foetus or during labour from recto-vaginally colonized women. The incidence of EOD in full-term new-borns has declined by approximately 90% in countries where there is routine screening of pregnant women for GBS recto-vaginal colonization at 35-37 weeks of gestational age and where IAP is provided 4 hours prior to delivery to colonized women. The strategy for routine screening for GBS colonization coupled with IAP, however, is not logistically feasible in most resource-constrained countries including Pakistan and has also been shown to be not cost-effective including in some high-income countries. The current CDC recommendation for the isolation of GBS from vaginal and rectal or recto-vaginal swabs is by initial growth in a selective broth medium with antibiotics, followed by subculture on blood agar or selective media.

This study aims to address the knowledge gaps to better inform the epidemiology of GBS in a low income setting and address some of the critical limitations of current data from low-middle income countries. Women who had normal vaginal delivery at term (>37 weeks of gestation age) will be enrolled in this study. Recto-vaginal swabs from the mothers will be collected for GBS.

All samples will be collected by trained midwives/physician before delivery. All newborns born to these mothers will be followed at 28th day after birth to assess their health status with emphasis on possible invasive disease episodes.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women age 13-49 years age.
* Pregnant women ≥37 weeks' gestation.
* Delivering by normal vaginal delivery.
* Are able to provide informed consent.

Exclusion Criteria:

1. Unwilling to consent to be on the study
2. Women who had taken any antibiotic treatment in previous two weeks 3 .Women who have blood transfusion in 30 days before delivery.

Ages: 13 Years to 49 Years | Sex: Female
Age Groups: Child, Adult
Gender Based: Yes — Pregnant women who are term delivery.
Study Population: This study will be focused on pregnant women who are delivered at term (≥37 weeks of gestation age). The study will be limited to women delivering by normal vaginal delivery. Gestational age staging will be determined by extrapolation of the date of last menstrual period and corroborated by physical examination of mother and/or infant and/or ultrasound report if available.
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of GBS colonization in pregnant women | 6-8 months
  i) Define the prevalence of GBS colonization in pregnant women at term-delivery and vertical acquisition thereof by the new-born in low income settlements in Karachi, Pakistan.

CONTACTS AND LOCATIONS:
Locations (1):
- PHC at Ibrahim Haidry Goth, Ali Akber Shah Colony, Rerhi Goth, Bhains Colony, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided